CLINICAL TRIAL: NCT01350141
Title: A Phase 2, Double-blind, Placebo-controlled, Randomized Study To Assess The Efficacy, Safety And Tolerability Of Pf-04950615 Following Multiple Intravenous Doses In Hypercholesterolemic Subjects On Maximum Dose Of Atorvastatin Or Rosuvastatin.
Brief Title: A Multiple Dose Study Of PF-04950615 (RN316) In Subjects On Maximum Doses Of Statins
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: B1481012
Record Dates: First submitted 2011-05-03; First posted 2011-05-09 (Estimated); Results first posted 2017-11-08 (Actual); Last update posted 2017-11-08 (Actual); Status verified 2017-10

CONDITIONS: Hypercholesterolemia; Dyslipidemia
Keywords: Hypercholesterolemia; dyslipidemia; high cholesterol; LDL; antibody; PCSK9; PF-04950615; RN316
MeSH Terms: conditions — Hypercholesterolemia; Dyslipidemias | interventions — bococizumab

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Treatment A (Placebo Comparator)
  Interventions: Other: Placebo
- Treatment B (Experimental)
  Interventions: Drug: PF-04950615 (RN316)
- Treatment C (Experimental)
  Interventions: Drug: PF-04950615 (RN316)

INTERVENTIONS:
Other: Placebo — An infusion lasting approximately 60 minutes
  Arms: Treatment A
Drug: PF-04950615 (RN316) — An infusion lasting approximately 60 minutes
  Arms: Treatment B
Drug: PF-04950615 (RN316) — An infusion lasting approximately 60 minutes
  Arms: Treatment C

SUMMARY:
PF-04950615 is a new investigational hypercholesterolemic agent that is being tested in this study to evaluate if it can lower LDL cholesterol.

ELIGIBILITY:
Inclusion Criteria:

* Body Mass Index (BMI) of 18.5 to 40 kg/m2
* On a stable maximum daily dose of a statin, defined as atorvastatin 80 mg or rosuvastatin 40 mg for a minimum of 45 days prior to Day 1.
* Lipids meet the following criteria twice during screening period:
* Fasting LDL C = or > 80 mg/dL;
* Fasting TG < 400 mg/dL.

Exclusion Criteria:

* History of a cardiovascular or cerebrovascular event or procedure (eg, MI, stroke, TIA, angioplasty) during the past year.
* Poorly controlled type 1 or type 2 diabetes mellitus.
* Poorly controlled hypertension.
* Fasting triglycerides > 400 mg/dL
* 12 lead ECG demonstrating QTcFF >455 msec at screening.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2011-06 (Actual); Primary Completion 2012-04 (Actual); Study Completion 2012-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (35):
- United States (29):
  - Achieve Clinical Research, LLC, Birmingham, Alabama
  - Advance Outcome Management, Inc., Garden Grove, California
  - Collaborative Neuroscience Network, Inc, Garden Grove, California
  - Collaborative Neuroscience Network, Inc., Long Beach, California
  - Elite Clinical Trials, Inc., Wildomar, California
  - Innovative Research of West Florida, Inc., Clearwater, Florida
  - Avail Clinical Research, LLC, DeLand, Florida
  - Kendall South Medical Center, Inc., Miami, Florida
  - Compass Research, LLC, Orlando, Florida
  - Atlanta Diabetes Associates, Atlanta, Georgia
  - Midwest Cardiology Associates, Overland Park, Kansas
  - Stark Pharmacy, Overland Park, Kansas
  - Vince and Associates Clinical Research, Overland Park, Kansas
  - Saint Luke's Hospital, Kansas City, Missouri
  - Saint Luke's Lipid and Diabetes Research Center, Kansas City, Missouri
  - Advance Clinical Research, St Louis, Missouri
  - Wake Internal Medicine Consultants, Inc., Raleigh, North Carolina
  - Wake Research Associates, LLC, Raleigh, North Carolina
  - Lynn Health Science Institute, Oklahoma City, Oklahoma
  - Oklahoma Cardiovascular Research Group, Oklahoma City, Oklahoma
  - Oklahoma Heart Hospital Physicians, Oklahoma City, Oklahoma
  - Oklahoma Heart Hospital, Oklahoma City, Oklahoma
  - Altoona Center for Clinical Research, Duncansville, Pennsylvania
  - DeGarmo Institute of Medical Research, Greer, South Carolina
  - Holston Medical Group, Kingsport, Tennessee
  - Texas Center for Drug Development, Inc, Houston, Texas
  - Martin Diagnostic Clinic, Tomball, Texas
  - Aspen Clinical Research, LLC, Orem, Utah
  - National Clinical Research - Richmond, Inc., Richmond, Virginia
- Canada (6):
  - The Medical Arts Health Research Group, Kelowna, British Columbia
  - Q & T Research Chicoutimi, Chicoutimi, Quebec
  - Centre de Recherche Clinique de Laval, Laval, Quebec
  - Diex Research Montreal Inc., Montreal, Quebec
  - Clinique des Maladies Lipidiques de Quebec Inc., Québec, Quebec
  - Diex Research Sherbrooke Inc., Sherbrooke, Quebec

REFERENCES:
- [Derived] Wang EQ, Kaila N, Plowchalk D, Gibiansky L, Yunis C, Sweeney K. Population PK/PD modeling of low-density lipoprotein cholesterol response in hypercholesterolemic participants following administration of bococizumab, a potent anti-PCSK9 monoclonal antibody. CPT Pharmacometrics Syst Pharmacol. 2023 Dec;12(12):2013-2026. doi: 10.1002/psp4.13050. Epub 2023 Nov 22. PMID 37994400
- [Derived] Wan H, Gumbiner B, Joh T, Riel T, Udata C, Forgues P, Garzone PD. Effects of Proprotein Convertase Subtilisin/Kexin Type 9 (PCSK9) Inhibition with Bococizumab on Lipoprotein Particles in Hypercholesterolemic Subjects. Clin Ther. 2017 Nov;39(11):2243-2259.e5. doi: 10.1016/j.clinthera.2017.09.009. Epub 2017 Oct 14. PMID 29037448
- [Derived] Udata C, Garzone PD, Gumbiner B, Joh T, Liang H, Liao KH, Williams JH, Meng X. A Mechanism-Based Pharmacokinetic/Pharmacodynamic Model for Bococizumab, a Humanized Monoclonal Antibody Against Proprotein Convertase Subtilisin/Kexin Type 9, and Its Application in Early Clinical Development. J Clin Pharmacol. 2017 Jul;57(7):855-864. doi: 10.1002/jcph.867. Epub 2017 Feb 9. PMID 28181260
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=B1481012&StudyName=A%20Multiple%20Dose%20Study%20Of%20PF-04950615%20%28RN316%29%20In%20Subjects%20On%20Maximum%20Doses%20Of%20Statins

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo: Participants received single intravenous infusion of placebo (normal saline) on Day 1, 29 and 57 along with atorvastatin 80 milligram (mg) tablet or rosuvastatin 40 mg tablet orally once daily from Day 1 to 141.
- PF-04950615 (RN316) 1 mg/kg: Participants received single intravenous infusion of PF-04950615 (RN316) 1 milligram per kilogram (mg/kg) on Day 1, 29 and 57 along with atorvastatin 80 mg tablet or rosuvastatin 40 mg tablet orally once daily from Day 1 to 141.
- PF-04950615 (RN316) 3 mg/kg: Participants received single intravenous infusion of PF-04950615 (RN316) 3 mg/kg on Day 1, 29 and 57 along with atorvastatin 80 mg tablet or rosuvastatin 40 mg tablet orally once daily from Day 1 to 141.
Period: Overall Study
Arm/Group | Placebo | PF-04950615 (RN316) 1 mg/kg | PF-04950615 (RN316) 3 mg/kg
Started | 15 | 15 | 16
Treated | 14 | 15 | 16
Completed | 12 | 15 | 15
Not Completed | 3 | 0 | 1
Not completed — Lost to Follow-up | 1 | 0 | 1
Not completed — Withdrawal by Subject | 1 | 0 | 0
Not completed — Randomized but not treated | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Safety analysis set included all participants who received at least 1 dose of study medication.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | PF-04950615 (RN316) 1 mg/kg | PF-04950615 (RN316) 3 mg/kg | Total
Number analyzed (Participants) | 14 | 15 | 16 | 45
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.1 (10.9) | 56.3 (10.9) | 57.6 (9.0) | 56 (10.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 7 | 9 | 22
  Male | 8 | 8 | 7 | 23

OUTCOME MEASURES:

1. Primary Outcome: Percent Change From Baseline in Low-density Lipoprotein Cholesterol (LDL-C) at Day 85
Description: Baseline value was calculated as the average of Day 7 and Day 1 measurements collected prior to study drug administration.
Time Frame: Baseline, Day 85
Population: Efficacy analysis set included all participants who received at least 1 dose of study medication and completed the Day 85 visit or dropped out prematurely, whichever was earlier. "Overall number of participants analyzed" signifies those participants who were evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Placebo | PF-04950615 (RN316) 1 mg/kg | PF-04950615 (RN316) 3 mg/kg
Number analyzed (Participants) | 12 | 15 | 14
percent change | 4.05 (21.688) | -14.95 (19.016) | -44.84 (27.186)
Statistical Analysis 1: Comparison: Placebo vs PF-04950615 (RN316) 1 mg/kg; Analysis was performed using analysis of covariance (ANCOVA) model with treatment, background statin as independent factors and treatment by background statin interaction, baseline LDL-C as covariate; Test type: Superiority or Other; p = 0.0137, ANCOVA; Least Squares (LS) Mean Difference = -21.81, 95% CI 2-sided [-38.85 to -4.77], Standard Error of Mean 8.385
Statistical Analysis 2: Comparison: Placebo vs PF-04950615 (RN316) 3 mg/kg; Analysis was performed using ANCOVA model with treatment, background statin as independent factors and treatment by background statin interaction, baseline LDL-C as covariate; Test type: Superiority or Other; p < 0.0001, ANCOVA; LS Mean Difference = -46.42, 95% CI 2-sided [-63.62 to -29.22], Standard Error of Mean 8.463

2. Secondary Outcome: Percentage of Participants Achieving Low-density Lipoprotein Cholesterol (LDL-C) Less Than 70 and Less Than 100 Milligram Per Deciliter (mg/dL)
Time Frame: Day 29, 57, 85
Population: Efficacy analysis set. "Overall number of participants analyzed" signifies those participants who were evaluable for this outcome measure and "Number of participants analyzed" signifies those participants who were evaluable for this measure at given time points, for each group respectively.
Measure: Number; unit: Percentage of participants
Arm/Group | Placebo | PF-04950615 (RN316) 1 mg/kg | PF-04950615 (RN316) 3 mg/kg
Number analyzed (Participants) | 13 | 15 | 16
Percentage of participants
  Day 29 less than 70 mg/dL: number analyzed (Participants) | 13 | 15 | 15
  Day 29 less than 70 mg/dL | 0.0 | 20.0 | 80.0
  Day 29 less than 100 mg/dL: number analyzed (Participants) | 13 | 15 | 15
  Day 29 less than 100 mg/dL | 15.4 | 86.7 | 100
  Day 57 less than 70 mg/dL: number analyzed (Participants) | 12 | 15 | 16
  Day 57 less than 70 mg/dL | 8.3 | 13.3 | 62.5
  Day 57 less than 100 mg/dL: number analyzed (Participants) | 12 | 15 | 16
  Day 57 less than 100 mg/dL | 33.3 | 73.3 | 87.5
  Day 85 less than 70 mg/dL: number analyzed (Participants) | 12 | 15 | 14
  Day 85 less than 70 mg/dL | 0.0 | 6.7 | 50.0
  Day 85 less than 100 mg/dL: number analyzed (Participants) | 12 | 15 | 14
  Day 85 less than 100 mg/dL | 33.3 | 73.3 | 92.9
Statistical Analysis 1: Comparison: Placebo vs PF-04950615 (RN316) 1 mg/kg; Day 29 less than 70 mg/dL: Analysis was performed using logistic regression with covariates baseline LDL-C and statin tested along with the treatment; Test type: Superiority or Other; p = 0.1900, Regression, Logistic; Odds Ratio (OR) = 7.825, 95% CI 2-sided [0.36 to 169.74]
Statistical Analysis 2: Comparison: Placebo vs PF-04950615 (RN316) 3 mg/kg; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.0057, Regression, Logistic; Odds Ratio (OR) = 72.518, 95% CI 2-sided [3.48 to 1512.10]
Statistical Analysis 3: Comparison: Placebo vs PF-04950615 (RN316) 1 mg/kg; Day 29 less than 100 mg/dL: Analysis was performed using logistic regression with covariates baseline LDL-C and statin tested along with the treatment; Test type: Superiority or Other; p = 0.0013, Regression, Logistic; Odds Ratio (OR) = 24.750, 95% CI 2-sided [3.49 to 175.63]
Statistical Analysis 4: Comparison: Placebo vs PF-04950615 (RN316) 3 mg/kg; [analysis description as in outcome 2, analysis 3]; Test type: Superiority or Other; p = 0.0006, Regression, Logistic; Odds Ratio (OR) = 47.326, 95% CI 2-sided [5.26 to 426.01]
Statistical Analysis 5: Comparison: Placebo vs PF-04950615 (RN316) 1 mg/kg; Day 57 less than 70 mg/dL: Analysis was performed using logistic regression with covariates baseline LDL-C and statin tested along with the treatment; Test type: Superiority or Other; p = 0.6611, Regression, Logistic; Odds Ratio (OR) = 1.635, 95% CI 2-sided [0.18 to 14.73]
Statistical Analysis 6: Comparison: Placebo vs PF-04950615 (RN316) 3 mg/kg; [analysis description as in outcome 2, analysis 5]; Test type: Superiority or Other; p = 0.0104, Regression, Logistic; Odds Ratio (OR) = 13.486, 95% CI 2-sided [1.84 to 98.61]
Statistical Analysis 7: Comparison: Placebo vs PF-04950615 (RN316) 1 mg/kg; Day 57 less than 100 mg/dL: Analysis was performed using logistic regression with covariates baseline LDL-C and statin tested along with the treatment; Test type: Superiority or Other; p = 0.0282, Regression, Logistic; Odds Ratio (OR) = 6.430, 95% CI 2-sided [1.22 to 33.89]
Statistical Analysis 8: Comparison: Placebo vs PF-04950615 (RN316) 3 mg/kg; [analysis description as in outcome 2, analysis 7]; Test type: Superiority or Other; p = 0.0042, Regression, Logistic; Odds Ratio (OR) = 15.257, 95% CI 2-sided [2.36 to 98.42]
Statistical Analysis 9: Comparison: Placebo vs PF-04950615 (RN316) 1 mg/kg; Day 85 less than 70 mg/dL: Analysis was performed using logistic regression with covariates baseline LDL-C and statin tested along with the treatment; Test type: Superiority or Other; p = 0.5164, Regression, Logistic; Odds Ratio (OR) = 2.967, 95% CI 2-sided [0.11 to 79.24]
Statistical Analysis 10: Comparison: Placebo vs PF-04950615 (RN316) 3 mg/kg; [analysis description as in outcome 2, analysis 9]; Test type: Superiority or Other; p = 0.0445, Regression, Logistic; Odds Ratio (OR) = 21.360, 95% CI 2-sided [1.08 to 422.94]
Statistical Analysis 11: Comparison: Placebo vs PF-04950615 (RN316) 1 mg/kg; Day 85 less than 100 mg/dL: Analysis was performed using logistic regression with covariates baseline LDL-C and statin tested along with the treatment; Test type: Superiority or Other; p = 0.0223, Regression, Logistic; Odds Ratio (OR) = 8.157, 95% CI 2-sided [1.35 to 49.37]
Statistical Analysis 12: Comparison: Placebo vs PF-04950615 (RN316) 3 mg/kg; [analysis description as in outcome 2, analysis 11]; Test type: Superiority or Other; p = 0.0070, Regression, Logistic; Odds Ratio (OR) = 13.587, 95% CI 2-sided [2.04 to 90.40]

3. Secondary Outcome: Percentage of Participants Achieving at Least 30 Percent Decrease in Low-density Lipoprotein Cholesterol (LDL-C)
Time Frame: Day 29, 57, 85
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | PF-04950615 (RN316) 1 mg/kg | PF-04950615 (RN316) 3 mg/kg
Number analyzed (Participants) | 13 | 15 | 16
percentage of participants
  Day 29: number analyzed (Participants) | 13 | 15 | 15
  Day 29 | 0.0 | 13.3 | 100
  Day 57: number analyzed (Participants) | 12 | 15 | 16
  Day 57 | 8.3 | 26.7 | 75.0
  Day 85: number analyzed (Participants) | 12 | 15 | 14
  Day 85 | 0.0 | 20.0 | 71.4
Statistical Analysis 1: Comparison: Placebo vs PF-04950615 (RN316) 1 mg/kg; Day 29: Analysis was performed using logistic regression with covariates baseline LDL-C and statin tested along with the treatment; Test type: Superiority or Other; p = 0.2928, Regression, Logistic; Odds Ratio (OR) = 5.647, 95% CI 2-sided [0.22 to 142.04]
Statistical Analysis 2: Comparison: Placebo vs PF-04950615 (RN316) 3 mg/kg; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p = 0.0014, Regression, Logistic; Odds Ratio (OR) = 591.174, 95% CI 2-sided [11.68 to 29922.99]
Statistical Analysis 3: Comparison: Placebo vs PF-04950615 (RN316) 1 mg/kg; Day 57: Analysis was performed using logistic regression with covariates baseline LDL-C and statin tested along with the treatment; Test type: Superiority or Other; p = 0.2339, Regression, Logistic; Odds Ratio (OR) = 3.468, 95% CI 2-sided [0.45 to 26.88]
Statistical Analysis 4: Comparison: Placebo vs PF-04950615 (RN316) 3 mg/kg; [analysis description as in outcome 3, analysis 3]; Test type: Superiority or Other; p = 0.0025, Regression, Logistic; Odds Ratio (OR) = 23.442, 95% CI 2-sided [3.03 to 181.11]
Statistical Analysis 5: Comparison: Placebo vs PF-04950615 (RN316) 1 mg/kg; Day 85: Analysis was performed using logistic regression with covariates baseline LDL-C and statin tested along with the treatment; Test type: Superiority or Other; p = 0.1786, Regression, Logistic; Odds Ratio (OR) = 8.502, 95% CI 2-sided [0.38 to 192.32]
Statistical Analysis 6: Comparison: Placebo vs PF-04950615 (RN316) 3 mg/kg; [analysis description as in outcome 3, analysis 5]; Test type: Superiority or Other; p = 0.0121, Regression, Logistic; Odds Ratio (OR) = 51.185, 95% CI 2-sided [2.37 to 1107.57]

4. Secondary Outcome: Change From Baseline in Lipid Parameters at Day 29, 57 and 85
Description: Lipid parameters included: high-density lipoprotein cholesterol (HDL-C), total cholesterol (TC), non-high-density lipoprotein-cholesterol (non-HDL-C), triglyceride (TG), apolipoprotein B (ApoB) and apolipoprotein A1 (ApoA1). Baseline value was calculated as the average of Day 7 and Day 1 measurements collected prior to study drug administration.
Time Frame: Baseline, Day 29, 57, 85
Population: Efficacy analysis set. 'Number of participants analyzed' = participants who were evaluable for this measure at given time points for each arm. Results for change at Day 85 for ApoB and ApoA1 were not reported as data was not collected for ApoB and ApoA1 at Day 85 due to an inadvertent omission in the protocol.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Placebo | PF-04950615 (RN316) 1 mg/kg | PF-04950615 (RN316) 3 mg/kg
Number analyzed (Participants) | 14 | 15 | 16
mg/dL
  Baseline HDL-C | 50.71 (12.277) | 50.63 (11.484) | 48.38 (12.905)
  Baseline TC | 191.14 (27.968) | 189.07 (26.443) | 195.34 (46.904)
  Baseline non-HDL-C | 140.43 (24.031) | 138.43 (29.850) | 146.97 (44.046)
  Baseline TG | 122.14 (56.077) | 156.50 (76.013) | 109.91 (45.854)
  Baseline ApoB | 91.57 (21.425) | 99.67 (21.784) | 100.88 (24.916)
  Baseline ApoA1 | 140.79 (25.057) | 146.73 (23.639) | 143.81 (31.503)
  Change at Day 29 HDL-C: number analyzed (Participants) | 13 | 15 | 15
  Change at Day 29 HDL-C | 0.92 (10.620) | -0.43 (4.330) | 5.53 (5.051)
  Change at Day 29 TC: number analyzed (Participants) | 13 | 15 | 15
  Change at Day 29 TC | 1.46 (20.821) | -23.00 (16.566) | -64.60 (22.634)
  Change at Day 29 non-HDL-C: number analyzed (Participants) | 13 | 15 | 15
  Change at Day 29 non-HDL-C | 0.54 (17.159) | -22.57 (16.804) | -71.40 (22.392)
  Change at Day 29 TG: number analyzed (Participants) | 13 | 15 | 15
  Change at Day 29 TG | -5.38 (42.455) | -23.37 (64.145) | -26.00 (39.128)
  Change at Day 29 ApoB: number analyzed (Participants) | 13 | 15 | 12
  Change at Day 29 ApoB | 6.77 (17.758) | -8.80 (14.561) | -43.75 (12.520)
  Change at Day 29 ApoA1: number analyzed (Participants) | 13 | 15 | 12
  Change at Day 29 ApoA1 | 6.15 (28.705) | -2.80 (17.350) | 8.58 (21.245)
  Change at Day 57 HDL-C: number analyzed (Participants) | 12 | 15 | 16
  Change at Day 57 HDL-C | -2.00 (7.138) | -0.23 (5.672) | 4.56 (8.072)
  Change at Day 57 TC: number analyzed (Participants) | 12 | 15 | 16
  Change at Day 57 TC | -12.79 (30.000) | -22.87 (33.173) | -52.66 (24.873)
  Change at Day 57 non-HDL-C: number analyzed (Participants) | 12 | 15 | 16
  Change at Day 57 non-HDL-C | -10.79 (31.447) | -22.63 (29.960) | -57.22 (29.026)
  Change at Day 57 TG: number analyzed (Participants) | 12 | 15 | 16
  Change at Day 57 TG | -5.88 (67.487) | -17.90 (44.184) | -23.97 (19.365)
  Change at Day 57 ApoB: number analyzed (Participants) | 12 | 15 | 15
  Change at Day 57 ApoB | 7.75 (22.483) | -8.47 (19.588) | -32.20 (20.772)
  Change at Day 57 ApoA1: number analyzed (Participants) | 13 | 15 | 15
  Change at Day 57 ApoA1 | 0.50 (23.240) | -1.27 (15.369) | 1.67 (21.043)
  Change at Day 85 HDL-C: number analyzed (Participants) | 12 | 15 | 14
  Change at Day 85 HDL-C | -1.42 (5.684) | 3.30 (6.959) | 1.79 (8.398)
  Change at Day 85 TC: number analyzed (Participants) | 12 | 15 | 15
  Change at Day 85 TC | 3.58 (26.618) | -17.60 (28.357) | -66.07 (45.818)
  Change at Day 85 non-HDL: number analyzed (Participants) | 12 | 15 | 14
  Change at Day 85 non-HDL | 5.00 (27.376) | -20.90 (25.716) | -64.32 (50.664)
  Change at Day 85 TG: number analyzed (Participants) | 12 | 15 | 15
  Change at Day 85 TG | 6.17 (48.767) | -21.10 (36.414) | -12.77 (41.558)

5. Secondary Outcome: Percent Change From Baseline in Lipid Parameters at Day 29, 57 and 85
Description: as for outcome 4
Time Frame: Baseline, Day 29, 57, 85
Population: Efficacy analysis set. "Number of participants analyzed" = participants who were evaluable for this measure at given time points for each arm. Results for percent change at Day 85 for ApoB and ApoA1 were not reported as data was not collected for ApoB and ApoA1 at Day 85 due to an inadvertent omission in the protocol.
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Placebo | PF-04950615 (RN316) 1 mg/kg | PF-04950615 (RN316) 3 mg/kg
Number analyzed (Participants) | 14 | 15 | 16
percent change
  Percent change at Day 29 HDL-C: number analyzed (Participants) | 13 | 15 | 15
  Percent change at Day 29 HDL-C | 0.50 (17.279) | -1.09 (7.935) | 11.93 (13.039)
  Percent change at Day 29 TC: number analyzed (Participants) | 13 | 15 | 15
  Percent change at Day 29 TC | 0.64 (10.318) | -12.63 (9.125) | -35.00 (13.281)
  Percent change at Day 29 non-HDL-C: number analyzed (Participants) | 13 | 15 | 15
  Percent change at Day 29 non-HDL-C | 0.74 (12.018) | -17.84 (14.222) | -52.65 (17.491)
  Percent change at Day 29 TG: number analyzed (Participants) | 13 | 15 | 15
  Percent change at Day 29 TG | 1.54 (38.088) | -11.15 (32.714) | -17.18 (23.596)
  Percent change at Day 29 ApoB: number analyzed (Participants) | 13 | 15 | 12
  Percent change at Day 29 ApoB | 11.65 (26.113) | -7.59 (13.739) | -43.43 (11.125)
  Percent change at Day 29 ApoA1: number analyzed (Participants) | 13 | 15 | 12
  Percent change at Day 29 ApoA1 | 5.63 (23.400) | -1.45 (10.716) | 8.34 (16.131)
  Percent change at Day 57 HDL-C: number analyzed (Participants) | 12 | 15 | 16
  Percent change at Day 57 HDL-C | -3.17 (14.071) | -0.80 (10.784) | 8.52 (15.458)
  Percent change at Day 57 TC: number analyzed (Participants) | 12 | 15 | 16
  Percent change at Day 57 TC | -7.69 (17.098) | -11.42 (16.477) | -26.58 (11.010)
  Percent change at Day 57 non-HDL-C: number analyzed (Participants) | 12 | 15 | 16
  Percent change at Day 57 non-HDL-C | -8.79 (23.929) | -14.74 (19.775) | -37.95 (15.373)
  Percent change at Day 57 TG: number analyzed (Participants) | 12 | 15 | 16
  Percent change at Day 57 TG | -3.94 (45.205) | -2.56 (33.634) | -20.56 (15.081)
  Percent change at Day 57 ApoB: number analyzed (Participants) | 12 | 15 | 15
  Percent change at Day 57 ApoB | 11.56 (25.094) | -7.03 (17.796) | -30.35 (17.065)
  Percent change at Day 57 ApoA1: number analyzed (Participants) | 12 | 15 | 15
  Percent change at Day 57 ApoA1 | 2.41 (19.469) | -0.02 (10.503) | 1.72 (15.505)
  Percent change at Day 85 HDL-C: number analyzed (Participants) | 12 | 15 | 14
  Percent change at Day 85 HDL-C | -1.75 (10.360) | 5.64 (12.221) | 3.18 (16.233)
  Percent change at Day 85 TC: number analyzed (Participants) | 12 | 15 | 15
  Percent change at Day 85 TC | 1.81 (13.580) | -9.36 (14.579) | -32.16 (20.664)
  Percent change at Day 85 non-HDL-C: number analyzed (Participants) | 12 | 15 | 14
  Percent change at Day 85 non-HDL-C | 3.28 (19.529) | -14.35 (17.206) | -40.37 (27.589)
  Percent change at Day 85 TG: number analyzed (Participants) | 12 | 15 | 15
  Percent change at Day 85 TG | 6.17 (36.703) | -8.28 (24.530) | -11.49 (32.647)

6. Secondary Outcome: Number of Participants With Treatment-Emergent Adverse Events (TEAEs)
Description: An adverse event (AE) was any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. Serious adverse event (SAE) was an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly. TEAEs are events between first dose of study drug and up to Day 141 that were absent before treatment or that worsened relative to pretreatment state. Treatment related: a TEAE deemed related to the study drug by the investigator. TEAEs included SAEs (TESAEs) as well as non-serious AEs which occurred during the study. The participants with TEAEs, TESAEs and treatment-related TEAEs were reported.
Time Frame: Day 1 up to Day 141
Population: Safety analysis set included all participants who received at least 1 dose of study medication.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | PF-04950615 (RN316) 1 mg/kg | PF-04950615 (RN316) 3 mg/kg
Number analyzed (Participants) | 14 | 15 | 16
Participants
  TEAEs (All causalities) | 9 | 12 | 9
  TESAEs (All causalities) | 0 | 1 | 0
  Treatment related TEAEs | 2 | 3 | 4

7. Secondary Outcome: Number of Treatment-Emergent Adverse Events (TEAEs) by Severity
Description: An AE was any untoward medical occurrence in participant who received study drug without regard to possibility of causal relationship. Investigator assessed adverse events as mild (does not interfere with participant's usual function), moderate (interferes to some extent with participant's usual function) or severe (interferes significantly with participant's usual function). All causality TEAEs were assessed for severity. TEAEs are events between first dose of study drug and up to Day 141 that were absent before treatment or that worsened relative to pretreatment state.
Time Frame: Day 1 up to Day 141
Population: Safety analysis set included all participants who received at least 1 dose of study medication.
Measure: Number; unit: Treatment-emergent AEs
Arm/Group | Placebo | PF-04950615 (RN316) 1 mg/kg | PF-04950615 (RN316) 3 mg/kg
Number analyzed (Participants) | 14 | 15 | 16
Treatment-emergent AEs
  Mild | 12 | 34 | 20
  Moderate | 2 | 19 | 7
  Severe | 0 | 0 | 0

8. Secondary Outcome: Number of Participants With Clinically Significant Laboratory Abnormalities
Description: Criteria for clinically significant laboratory abnormalities were based on investigator's discretion. Total number of participants who met the criteria for any laboratory abnormal findings were reported. Laboratory parameters included: hematology, coagulation, liver function, renal function, electrolytes, hormones, chemistry and urinalysis. Screening was 21 days prior to start of study treatment.
Time Frame: Screening up to Day 141
Population: Safety analysis set included all participants who received at least 1 dose of study medication.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | PF-04950615 (RN316) 1 mg/kg | PF-04950615 (RN316) 3 mg/kg
Number analyzed (Participants) | 14 | 15 | 16
Participants | 12 | 15 | 16

9. Secondary Outcome: Number of Participants With Clinically Significant Changes in Vital Signs and Electrocardiogram (ECG) Parameters
Description: Number of participants with clinically significant changes in vital signs and ECG findings were reported. Criteria for clinical significant vital signs: maximum increase or decrease from baseline in supine systolic blood pressure (BP) greater than or equal to (>=) 30 millimeter of mercury (mmHg), maximum increase or decrease from baseline in supine diastolic BP of >=20 mmHg. Criteria for clinically significant ECG parameters: maximum increase of >=25 percent (%) for baseline value of greater than 200 millisecond (msec) or maximum increase of >=50% for baseline value of less than or equal to (<=) 200 msec for PR and QRS interval, maximum increase from baseline of greater than (>) 30 to <=60 msec and maximum increase from baseline of >60 msec for QT interval corrected using the Fridericia's formula (QTCF). Screening was 21 days prior to start of study treatment.
Time Frame: Screening up to Day 141
Population: Safety analysis set included all participants who received at least 1 dose of study medication.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | PF-04950615 (RN316) 1 mg/kg | PF-04950615 (RN316) 3 mg/kg
Number analyzed (Participants) | 14 | 15 | 16
Participants
  Supine systolic BP: Maximum increase >=30mmHg | 0 | 2 | 2
  Supine diastolic BP: Maximum increase >=20mmHg | 2 | 0 | 3
  Supine systolic BP: Maximum decrease >=30mmHg | 1 | 3 | 3
  Supine diastolic BP: Maximum decrease >=20mmHg | 2 | 4 | 1
  PR interval: >=25/50% increase | 0 | 0 | 0
  QRS interval: >=25/50% increase | 0 | 0 | 0
  QTCF: Maximum increase >30 to <=60 msec | 3 | 1 | 1
  QTCF: Maximum increase >60 msec | 0 | 0 | 0

10. Secondary Outcome: Number of Participants With Anti-drug (Anti-PF-04950615) Antibody (ADA)
Description: Human serum samples of participants who received PF-04950615 (RN316) were analyzed for the presence of anti-PF-04950615 antibodies by using the semi quantitative enzyme-linked immunosorbent assay (ELISA). Results with titer value >=4.32 nanogram per milliliter of anti-PF-04950615 antibodies were counted as positive. Number of participants with presence of anti-PF-04950615 antibodies were reported in this outcome measure.
Time Frame: Day 1 up to Day 141
Population: Analysis set included all participants who received at least 1 dose of PF-04950615 (RN316).
Measure: Number; unit: participants
Arm/Group | PF-04950615 (RN316) 1 mg/kg | PF-04950615 (RN316) 3 mg/kg
Number analyzed (Participants) | 15 | 16
participants | 0 | 0

ADVERSE EVENTS:
Description: The same event may appear as both an AE and a SAE. However, what is presented are distinct events. An event may be categorized as serious in one participant and as nonserious in another participant, or one participant may have experienced both a serious and nonserious event during the study. Safety population.
Arm/Group | Placebo | PF-04950615 (RN316) 1 mg/kg | PF-04950615 (RN316) 3 mg/kg
Serious Adverse Events (participants affected / at risk) | 0/14 | 1/15 | 0/16
Other Adverse Events (participants affected / at risk) | 9/14 | 12/15 | 9/16
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=14) | PF-04950615 (RN316) 1 mg/kg (N=15) | PF-04950615 (RN316) 3 mg/kg (N=16)
Non-cardiac chest pain (General disorders) | 0 | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=14) | PF-04950615 (RN316) 1 mg/kg (N=15) | PF-04950615 (RN316) 3 mg/kg (N=16)
Atrioventricular block first degree (Cardiac disorders) | 0 | 0 | 1
Sinus bradycardia (Cardiac disorders) | 0 | 1 | 0
Tachycardia (Cardiac disorders) | 0 | 1 | 0
Conjunctival haemorrhage (Eye disorders) | 0 | 1 | 0
Conjunctivitis allergic (Eye disorders) | 0 | 1 | 0
Vision blurred (Eye disorders) | 0 | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 1
Abdominal pain upper (Gastrointestinal disorders) | 0 | 1 | 0
Colitis microscopic (Gastrointestinal disorders) | 0 | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 0 | 2
Flatulence (Gastrointestinal disorders) | 0 | 1 | 0
Nausea (Gastrointestinal disorders) | 0 | 3 | 0
Oral pain (Gastrointestinal disorders) | 0 | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 0 | 1
Axillary pain (General disorders) | 0 | 1 | 0
Fatigue (General disorders) | 0 | 1 | 0
Non-cardiac chest pain (General disorders) | 0 | 2 | 0
Oedema peripheral (General disorders) | 1 | 0 | 0
Abscess (Infections and infestations) | 0 | 1 | 0
Abscess limb (Infections and infestations) | 0 | 1 | 0
Cellulitis (Infections and infestations) | 0 | 0 | 1
Gastroenteritis (Infections and infestations) | 0 | 1 | 0
Herpes zoster (Infections and infestations) | 0 | 0 | 1
Influenza (Infections and infestations) | 0 | 0 | 1
Nasopharyngitis (Infections and infestations) | 1 | 1 | 1
Oral herpes (Infections and infestations) | 1 | 0 | 0
Sinusitis (Infections and infestations) | 0 | 1 | 0
Tooth abscess (Infections and infestations) | 0 | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 4 | 1
Joint dislocation (Injury, poisoning and procedural complications) | 0 | 0 | 1
Joint injury (Injury, poisoning and procedural complications) | 0 | 1 | 1
Muscle strain (Injury, poisoning and procedural complications) | 0 | 1 | 0
Road traffic accident (Injury, poisoning and procedural complications) | 0 | 1 | 0
Blood cortisol decreased (Investigations) | 1 | 1 | 0
Blood creatinine increased (Investigations) | 0 | 1 | 0
Hyperuricaemia (Metabolism and nutrition disorders) | 0 | 1 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 1 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Jaw cyst (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Joint stiffness (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Dizziness (Nervous system disorders) | 0 | 1 | 0
Dysgeusia (Nervous system disorders) | 1 | 1 | 0
Essential tremor (Nervous system disorders) | 0 | 1 | 0
Headache (Nervous system disorders) | 3 | 3 | 3
Hypoaesthesia (Nervous system disorders) | 1 | 0 | 0
Neuralgic amyotrophy (Nervous system disorders) | 1 | 0 | 0
Paraesthesia (Nervous system disorders) | 0 | 1 | 0
Nocturia (Renal and urinary disorders) | 0 | 1 | 0
Breast tenderness (Reproductive system and breast disorders) | 0 | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Acne (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Exfoliative rash (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Skin fissures (Skin and subcutaneous tissue disorders) | 0 | 0 | 1

LIMITATIONS AND CAVEATS:
Due to an inadvertent omission in the protocol at Day 85, presented limitations in data collection and the assessment of treatment effect on ApoA1 and ApoB for Day 85.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.